CLINICAL TRIAL: NCT06616896
Title: Precision Rehabilitation: Mechanisms and Efficacy of Vibration in Exercise Training for Degenerative Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 202404060RIND
Record Dates: First submitted 2024-09-18; First posted 2024-09-27 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthristis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continued mode vibration intervention (Experimental)
  Interventions: Device: vibration
- Pause mode vibration intervention (Experimental)
  Interventions: Device: vibration

INTERVENTIONS:
Device: vibration — Each participant will randomly receive four different vibration conditions (2 frequencies × 2 vibration modes = 4 conditions) in a different order. Considering that the current research range of local vibration frequency is 10 to 150 Hz the frequencies with low and high frequencies (30/60Hz) will be selected. The location chosen for this study is the quadriceps muscle belly. Two-minute vibrations will improve muscle strength without any fatigue side effects. Two vibration modes include providing a two-minute continuous vibration intervention and only providing vibration during the rest position before executing the functional test.

SUMMARY:
Knee osteoarthritis (OA) is a common degenerative disease in older populations. Chronic pain, quadriceps weakness, limited daily activities, lack of mobility, and balance and walking dysfunction are the most common symptoms. The overall aim of this study is to employ artificial intelligence (AI) based on the concepts of precision rehabilitation to design a wearable multifunctional vibration knee brace that is best suited for improving degenerative knee OA in functional performance and pain relief. The investigators hypothesize that this AI-based precision rehabilitation device will improve the functional performance and pain relief of elderly patients with degenerative knee OA compared to conventional treatments. The expected outcome of this proposed study will be evidence of the feasibility and efficacy of exercise training combined with vibration intervention using an AI knee brace in patients with knee OA. This four-year study will achieve the following three specific aims:

Aim 1: To identify the optimal mode of vibration intervention during functional movements in patients with knee OA.

Patients with knee OA will be recruited and receive different vibration conditions at the thigh muscles during functional movements. This cross-sectional, single-blind, randomized study will provide reference values based on the results of hemodynamics in the brain and the local muscles, as well as muscle strength tests to determine the best vibration intervention mode for patients with knee OA. The investigators will recruit 60 patients with knee OA and assess changes in hemodynamics, proprioception, functional performance, and muscle strength performance pre- and post-vibration. The optimized vibration intervention mode of this study will contribute to the reference foundation for vibration intervention in patients with knee OA, as well as the implementation decision-making of aims 2 and 3 of this study.

Aim 2: To develop an AI knee brace that can be used as a clinical evaluation tool and implement vibration intervention at the right time.

The investigators will develop an AI knee brace that can collect movement data, such as kinematics, kinetics, and muscle activities, as inputs. Then, it outputs computed data such as functional task recognition and joint force estimation. Using AI algorithms, the investigators will analyze the biomechanical data collected by the sensors embedded in the knee brace and adjust the vibration frequency, intensity, and duration to optimize the therapeutic effects. This study will recruit 10 patients with knee OA and 10 age-matched healthy elderly participants. The AI knee brace will be validated for its evaluation function and therapeutic effects.

Aim 3: To determine the effects of exercise training combined with vibration intervention using the AI knee brace in patients with knee OA.

The investigators used sealed letter to conduct a randomized control trial (RCT), using the developed AI knee brace in conjunction with exercise training to enhance functional performance and relieve pain in patients with knee OA. This exercise training can integrate real-time knee motion assistance and muscle activity feedback, which will help patients control the knee while exercising to avoid sports injuries. The 60 knee OA patients will be randomly assigned into two groups. The experimental group will receive a combined AI knee brace and exercise training intervention for 8 weeks, while the control group will receive standard exercise training alone. Hemodynamic and biomechanical analyses will determine the outcome at four-time points (i.e., pre-training, post-training, 3-month post-training, and 1-year post-training).

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 to 80 years
* A diagnosis of knee OA (Kellgren and Lawrence grade 1~3 on X-ray) according to the American College of Rheumatology's criteria.

Exclusion Criteria:

* Knee or hip surgery
* Systemic arthritis
* Neurological disorders.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
muscle strength | Muscle strength outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  muscle strength will be measured by maximal voluntary isometric contraction (MVIC) of the knee extension using a dynamometer muscle tester. All muscle strength data will be normalized with body weight.
Muscle activity | Muscle activity outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Muscle activity will be collected by electrography (EMG). Electrode sites (quadriceps) will be shaved and cleaned with alcohol to enhance signal quality. All electrodes were placed longitudinally over the muscle.
Proprioception | Proprioception outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Knee joint position sense absolute error will be measured using Inertial Measurement Unit (IMU) before and after vibration intervention to evaluate proprioception. IMU is a device that measures and reports an object's specific force, angular rate, and sometimes magnetic field surrounding the body using a combination of sensors, including accelerometers, gyroscopes, and sometimes magnetometers.
Hemodynamics analysis of Oxygenated Hemoglobin | Oxygenated Hemoglobin outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Hemodynamics analysis of Oxygenated Hemoglobin will focus on quadriceps muscles and cerebral hemodynamics data and will be monitored simultaneously using fNIRS during vibration. The areas of interest in cerebral hemodynamics mainly focus on the dorsal medial prefrontal cortex (DMPFC) because DMPFC plays an essential role in rapid error prediction. The investigators will conduct data analysis by comparing the changes in parameters of Oxygenated Hemoglobin before and after vibration intervention.
Hemodynamics analysis of Deoxygenated Hemoglobin | Deoxygenated Hemoglobin outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Hemodynamics analysis of Deoxygenated Hemoglobin will focus on quadriceps muscles and cerebral hemodynamics data and will be monitored simultaneously using fNIRS during vibration. The areas of interest in cerebral hemodynamics mainly focus on the dorsal medial prefrontal cortex (DMPFC) because DMPFC plays an essential role in rapid error prediction. The investigators will conduct data analysis by comparing the changes in parameters of Deoxygenated Hemoglobin before and after vibration intervention.
Hemodynamics analysis of Total Hemoglobin | Total Hemoglobin outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Hemodynamics analysis of Total Hemoglobin will focus on quadriceps muscles and cerebral hemodynamics data and will be monitored simultaneously using fNIRS during vibration. The areas of interest in cerebral hemodynamics mainly focus on the dorsal medial prefrontal cortex (DMPFC) because DMPFC plays an essential role in rapid error prediction. The investigators will conduct data analysis by comparing the changes in parameters of Oxygenated Hemoglobin before and after vibration intervention.

SECONDARY OUTCOMES:
Five-sit-to-stand tests(5-STS) | Five-sit-to-stand tests(5-STS) outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Functional movement assessment will be assessed through Five-sit-to-stand tests(5-STS)
Time up and go test (TUG) | Time up and go test (TUG) outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Functional movement assessment will be assessed through Time up and go test (TUG)
10-meter walking test | 10-meter walking test outcome measure will be assessed immediately after vibration and will be reported through study completion, an average of 1 year
  Functional movement assessment will be assessed through 10-meter walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital International Medical Service Center, Taipei, Taiwan